CLINICAL TRIAL: NCT00996190
Title: Study to Determine the Best Regimen for Administration of Phenylephrine During Spinal Anesthesia for Cesarean Delivery, as Determined by Maternal Blood Pressure and Cardiac Output
Brief Title: Best Regimen for Phenylephrine Administration During Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose Carvalho, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-03
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Cesarean Section; Cardiac Output; Hypotension
Keywords: transthoracic bioreactance; noninvasive monitoring; vasopressor; blood pressure
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenylephrine Intermittent Bolus (Active Comparator): Bolus syringe will contain 120 micrograms/mL of phenylephrine. Infusion solution bag will contain placebo (saline solution).
  Interventions: Drug: Phenylephrine
- Phenylephrine Continuous Infusion (Active Comparator): Infusion solution bag will contain 120 micrograms/mL of phenylephrine. Bolus syringe will contain placebo (saline solution).
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine — phenylephrine 120 micrograms/mL, administered either by continuous infusion or by intermittent bolus dose

SUMMARY:
During Cesarean delivery, phenylephrine is used to maintain the patient's blood pressure. Low blood pressure is the most common side effect of the spinal medication used to anesthetize the patient prior to the start of surgery. This low blood pressure can also trigger unpleasant side effects such as nausea, vomiting and low Apgar scores for the baby.

Currently there are 2 methods of phenylephrine administration during Cesarean section. One method is by intermittent bolus and the other is by continuous infusion. It is ideal to have a regimen for phenylephrine administration that maintains blood pressure without compromising cardiac output.

In this study, cardiac output and blood pressure will be measured by transthoracic bioimpedance, which is a new technique of noninvasive continuous cardiac output monitoring.

The hypothesis of this study is that the continuous infusion of phenylephrine will be equally effective in maintaining blood pressure as compared to the intermittent injection, and will induce less hemodynamic changes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to communicate in English
* Elective Cesarean Delivery under spinal anesthesia
* Normal singleton pregnancy beyond 36 weeks gestation
* ASA physical status I/II
* Weight 50-100 kg, height 150-180 cm
* Age over 18 years

Exclusion Criteria:

* Patient refusal
* Inability to communicate in English
* Allergy or hypersensitivity to phenylephrine
* Preexisting or pregnancy-induced hypertension
* Cardiovascular or cerebrovascular disease
* Fetal abnormalities
* History of diabetes, excluding gestational diabetes
* Contra-indications for spinal anesthesia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The maximum decrease in cardiac output in the pre-delivery period. | 30 minutes

SECONDARY OUTCOMES:
Maximum decrease in heart rate in the pre-delivery period. | 30 minutes
Incidence of hypotension in the pre-delivery period (BP < 80% baseline) | 30 minutes
Incidence of hypertension in the pre-delivery period (BP > 120% baseline) | 30 minutes
Incidence of nausea and vomiting in the pre-delivery period | 30 minutes
Total dose of phenylephrine in the pre-delivery period | 30 minutes
Umbilical artery and vein blood gases | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada